CLINICAL TRIAL: NCT00095420
Title: Peer Related School Interventions in Autism
Brief Title: Relationship Training for Children With Autism and Their Peers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: U54MH068172 (NIH); U54MH068172 (NIH); DDTR BD-DD
Record Dates: First submitted 2004-11-04; First posted 2004-11-05 (Estimated); Last update posted 2025-10-30 (Actual); Status verified 2022-02

CONDITIONS: Autism; Autistic Disorder
Keywords: Interpersonal Relationships; Child
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Participants with autism will receive social skills training targeting children with autism
  Interventions: Behavioral: Social skills training targeting children with autism
- 2 (Experimental): Participants without autism will receive social skills training to increase acceptance of peers with autism
  Interventions: Behavioral: Social skills training of peers without autism
- 3 (Experimental): Participants with and without autism will receive a combination treatment of social skills/education about autism
  Interventions: Behavioral: Combination treatment of social skills/education about autism
- 4 (Active Comparator): Participants with and without autism will receive usual training provided by their school district
  Interventions: Behavioral: Usual training

INTERVENTIONS:
Behavioral: Social skills training targeting children with autism — Sessions will focus on improving the social skills of autistic children. Thirty-minute sessions will be held twice a week for 6 weeks.
  Arms: 1
Behavioral: Social skills training of peers without autism — Sessions will involve educating the peers of autistic children to increase their acceptance of their autistic peers. Thirty-minute sessions will be held twice a week for 6 weeks.
  Arms: 2
Behavioral: Combination treatment of social skills/education about autism — The combination treatment includes children with and without autism. Sessions will involve social skills training and education about autism to increase acceptance of autistic peers. Training will be conducted twice a week for 6 weeks
  Arms: 3
Behavioral: Usual training — Participants will receive the usual training offered in their local school districts.
  Arms: 4

SUMMARY:
This study will determine whether peer interaction training interventions are effective in enhancing the social relationships of children with autism.

DETAILED DESCRIPTION:
Children with autism often have poor relationships with other children during their childhood and through their adult lives. A number of peer-related intervention models have been developed, but these models have not been thoroughly reviewed or implemented within the school setting. This study will examine the social inclusion of children with autism, following different peer-related interventions training children with autism and their peers.

Children will be randomly assigned to one of four interventions that comprise all autistic children, all nonautistic children, or a mixed group of both. The first intervention focuses on improving the social skills of autistic children. The second intervention involves educating the peers of autistic children to increase their acceptance of their autistic peers. The third intervention is a combination of the first two interventions. Children assigned to the fourth intervention will receive the usual training offered in their local school districts. Training for each group will be conducted twice a week for 6 weeks.

Characteristics of the autistic child will be assessed through an interview that evaluates intelligence quotient (IQ), language skills, and social interaction. Teachers will be asked to complete a questionnaire describing the autistic child and his or her interaction with peers. The autistic children will complete a friendship survey, clinical global impressions scales, and a battery of neuropsychiatric tests. All assessments will be conducted at study start and again at study completion.

ELIGIBILITY:
Inclusion Criteria for Autistic and Nonautistic Participants:

* Autistic OR nonautistic peer of autistic child
* Full inclusion in a classroom with nonautistic children
* Currently in kindergarten or grades 1 through 5
* Intelligence quotient higher than 70
* Expectation to stay in the same school and classroom for the duration of the study
* Able to provide parent consent and child assent

Exclusion Criteria:

* Mental age-equivalent less than 4 years
* Conditions other than autism, or sensory or motor impairments

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2003-09; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Social network involvement of autistic children | Measured before and after treatment and at 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Marian Sigman, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Anderson A, Locke J, Kretzmann M, Kasari C; AIR-B Network. Social network analysis of children with autism spectrum disorder: Predictors of fragmentation and connectivity in elementary school classrooms. Autism. 2016 Aug;20(6):700-9. doi: 10.1177/1362361315603568. Epub 2015 Nov 13. PMID 26567264
- [Derived] Locke J, Shih W, Kretzmann M, Kasari C. Examining playground engagement between elementary school children with and without autism spectrum disorder. Autism. 2016 Aug;20(6):653-62. doi: 10.1177/1362361315599468. Epub 2015 Sep 4. PMID 26341991
- [Derived] Dean M, Kasari C, Shih W, Frankel F, Whitney R, Landa R, Lord C, Orlich F, King B, Harwood R. The peer relationships of girls with ASD at school: comparison to boys and girls with and without ASD. J Child Psychol Psychiatry. 2014 Nov;55(11):1218-25. doi: 10.1111/jcpp.12242. Epub 2014 Jul 16. PMID 25039696
- [Derived] Locke J, Rotheram-Fuller E, Kasari C. Exploring the social impact of being a typical peer model for included children with autism spectrum disorder. J Autism Dev Disord. 2012 Sep;42(9):1895-905. doi: 10.1007/s10803-011-1437-0. PMID 22215436
- [Derived] Kasari C, Rotheram-Fuller E, Locke J, Gulsrud A. Making the connection: randomized controlled trial of social skills at school for children with autism spectrum disorders. J Child Psychol Psychiatry. 2012 Apr;53(4):431-9. doi: 10.1111/j.1469-7610.2011.02493.x. Epub 2011 Nov 26. PMID 22118062
- See also: Click here for more information about this study and others at the University of California, Los Angeles Center for Autism Research and Treatment Web site. — http://www.semel.ucla.edu/autism
- Available data/document: Clinical Study Report — http://pubmed.ncbi.nlm.nih.gov/22118062/
- Available data/document: Clinical Study Report — http://www.researchgate.net/publication/10751612_General_Education_Teacher
- Available data/document: Clinical Study Report — http://pubmed.ncbi.nlm.nih.gov/20673234/
- Available data/document: Clinical Study Report — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3076578/
- Available data/document: Clinical Study Report — http://pubmed.ncbi.nlm.nih.gov/27620949/